CLINICAL TRIAL: NCT05543720
Title: Nurse-led Integrated Care of Complex Patients Facilitated By Telemonitoring: The Safe, Managed, and Responsive Transitions (SMaRT) Study
Brief Title: Evaluation of Nurse-led Integrated Care of Complex Patients Facilitated By Telemonitoring: The SMaRT Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Markham Stouffville Hospital (Other); William Osler Health System (Other); Health Sciences North (Other); Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-5835; 510037 (Other Grant/Funding Number: CIHR); SMaRT Study (Other: UHN)
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure，Congestive; Mental Health (Depression); Diabetes Mellitus; Chronic Obstructive Pulmonary Disease; Hypertension
Keywords: Telemonitoring; Smartphone application; Chronic disease management; Remote monitoring; Multiple chronic conditions; mHealth; Nurse-led; Holistic care
MeSH Terms: conditions — Heart Failure; Psychological Well-Being; Depression; Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive; Hypertension; Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: Propensity-score matched controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control groups will be compared to 350 patients who received standard of care via propensity-matched controls from the ICES provincial database.
- Telemonitoring (Medly MCC) (Experimental): Medly is a smartphone application allows patients with heart failure, diabetes, depression, hypertension, and/or COPD to measure and record their daily self-reported symptoms. This monitoring information is then transmitted wirelessly to a data server where an algorithm is used to generate an alert to a healthcare provider as necessary. The patient also receives an automated self-care message based on their measurements and reported symptoms.
  Interventions: Device: Medly

INTERVENTIONS:
Device: Medly — Medly will enable patients with HF, COPD, Hypertension, Mental Health, or Diabetes to input measurements with wireless home medical devices and to answer symptom questions on the smartphone. The measurements will be automatically and wirelessly transmitted to the mobile phone and then to a data server. Automated self-care instructions/messages will be sent to the patient based on the readings and reported symptoms. If there are signs of their status deteriorating, an alert will be sent to a clinician that is responsible for the particular chronic condition of concern. The clinicians will have all the relevant patient data sent to them and will be able to access (through a secure web portal) to view historical and trending data for their patients.
  Arms: Telemonitoring (Medly MCC)

SUMMARY:
In Canada, 3 out of 4 Canadians aged 65 and older have at least one chronic condition, while 1 in 4 seniors reported having three or more. Caring for complex patients who usually have multiple chronic conditions (MCC) is one of the biggest challenges facing our healthcare system. For patients, the lack of coordination and continuity of care as they transfer between healthcare settings and healthcare providers (HCPs) often results in a higher risk of readmission, suboptimal and fragmented care plans, delays in required medical intervention, inadequate self-care, and confusion on whom they should contact when they have questions. For the patient's care team, they often have no indication how patients are doing between clinic visits unless the patient can provide a log of their home measurements (e.g., blood pressure). Therefore, they are unable to detect and intervene if their patient's health is worsening between visits.

In order to address this increasing need to bridge the current gap in clinical management and self-care of complex patients during their transition from healthcare settings to home care, our team aims to design, implement and evaluate the SMaRT (Safe, Managed, and Responsive Transitions) Clinic, a nurse-led integrated care model facilitated by telemonitoring (TM). Specifically, the SMaRT Clinics aim to meaningfully introduce a nurse (or nurse practitioner) role to improve clinical coordination across patient care teams and reinforce proper self-care education through the use of telemonitoring. This project will be conducted in two phases across four years; Phase I: Design and Development, and Phase II: Implementation and Effectiveness Evaluation. Phase II research activities include enrolling 350 patients with complex chronic conditions in the SMaRT clinics across four study sites. The implementation and effectiveness of the SMaRT clinics will be evaluated through a mix of semi-structured interviews, ethnographic observation, patient questionnaires, and analyses of health utilization outcomes using propensity-matched controls from the ICES provincial database.

DETAILED DESCRIPTION:
The overall objective of this study is to design, implement, and evaluate SMaRT Clinics at four hospitals across Ontario serving complex patients transitioning home from the hospital in urban, suburban and rural settings. Instead of developing new technology for the nurse-led SMaRT Clinic, an existing validated TM system that is able to monitor patients with multiple chronic conditions, named Medly, was chosen. Medly was developed at eHealth Innovation (now called the Centre for Digital Therapeutics), UHN and was designed to monitor a medley of chronic conditions, and has been evaluated in trials for single chronic conditions and multiple chronic conditions. For the purposes of this trial, Medly will enable the TM of heart failure, COPD, diabetes, hypertension, and depression.

The patient-facing technology includes the Medly smartphone application (app). The app enables patients to complete symptom surveys and record physiological measures using peripheral devices relevant to their chronic condition (e.g., weight scale, blood pressure monitor, and/or blood glucose monitoring). Designed as a modular app, features and parameters to be monitored can be added and removed, and target values for each parameter (e.g. blood pressure) can be individualized according to the needs of each patient. The inputted measures are processed by an embedded rules-based algorithm (customized to the patient by the setting of target thresholds) which triggers appropriate self-care messages being displayed to the patient within the app (e.g., instructing patients to take their prescribed medication, informing patients to contact their care team, etc.). Other features of the Medly app include the ability to view a historical record of their inputted readings, view graphical trends of blood glucose and blood pressure values, and to assist with adherence, an automated phone call to remind patients if they have not yet taken their readings by the appropriate time for their condition.

The clinician-facing technology includes the Medly dashboard. To support clinical decision-making, clinicians are alerted to clinically significant changes to patient health status and are able to assess alerts generated by the embedded algorithm and review patient data, including which parameters triggered the alert, prescribed medications, graphical trends of lab results and relevant measures, and contact information. Clinicians may also be informed of triggered alerts through email notifications. Information presented on the Medly dashboard may be leveraged to inform clinical decision-making throughout the patient's follow-up care journey.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Discharged from hospital or seen within 48 hours of discharge at Health Sciences North (HSN), William Osler Health Systems (WOHS), Women's College Hospital (WCH), and Markham Stouffville Hospital (MSH).
3. Have at least one complex chronic condition (i.e., heart failure, complex obstructive pulmonary disease (COPD), hypertension, diabetes, and/or depression) that would benefit if monitored through telemonitoring.
4. Able to comply with use of the telemonitoring application and applicable peripheral devices (e.g., able to stand on the weight scale, able to answer symptom questions, etc.)
5. Able to read, write and speak English or have a caregiver who is able to do so on their behalf.
6. Patients must have been discharged from hospital within 2 weeks during their recruitment into the study (or will be recruited prior to their discharge).

Exclusion Criteria:

1. Patients who are discharged from hospital with the intent to be admitted to a long-term care facility will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Death and/or all-cause unplanned readmission | 30 days
  The primary outcome measure for effectiveness evaluation will be a composite of death and all-cause unplanned readmission over 30 days.

SECONDARY OUTCOMES:
Death and/or all-cause unplanned readmission | 6 months and at 1-year
  The secondary outcome measure for effectiveness evaluation will be a composite of death and all-cause unplanned readmission over 6 months and 1 year.
All-cause mortality | Over 30 days, at 6 months, and at 1-year follow-up
  All-cause mortality
Readmissions | Over 30 days, at 6 months, and at 1-year follow-up
  The number of Readmissions to Hospital
Days alive and out-of-hospital | Over 30 days, at 6 months, and at 1-year follow-up
  Days alive and out-of-hospital

CONTACTS AND LOCATIONS:
Overall Officials: Emily Seto, PhD, Principal Investigator — University of Toronto
Locations (4):
- Canada (4):
  - William Osler Health System, Brampton, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - Oak Valley Health Hospital, Markham, Ontario
  - Women's College Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Spall HGC, Rahman T, Mytton O, Ramasundarahettige C, Ibrahim Q, Kabali C, Coppens M, Brian Haynes R, Connolly S. Comparative effectiveness of transitional care services in patients discharged from the hospital with heart failure: a systematic review and network meta-analysis. Eur J Heart Fail. 2017 Nov;19(11):1427-1443. doi: 10.1002/ejhf.765. Epub 2017 Feb 24. PMID 28233442
- [Background] Haggerty JL, Reid RJ, Freeman GK, Starfield BH, Adair CE, McKendry R. Continuity of care: a multidisciplinary review. BMJ. 2003 Nov 22;327(7425):1219-21. doi: 10.1136/bmj.327.7425.1219. PMID 14630762
- [Background] Seto E, Leonard KJ, Cafazzo JA, Masino C, Barnsley J, Ross HJ. Self-care and quality of life of heart failure patients at a multidisciplinary heart function clinic. J Cardiovasc Nurs. 2011 Sep-Oct;26(5):377-85. doi: 10.1097/JCN.0b013e31820612b8. PMID 21263339
- [Background] Liddy C, Blazkho V, Mill K. Challenges of self-management when living with multiple chronic conditions: systematic review of the qualitative literature. Can Fam Physician. 2014 Dec;60(12):1123-33. PMID 25642490
- [Background] Gordon K, Gray CS, Dainty KN, deLacy J, Seto E. Nurse-Led Models of Care for Patients with Complex Chronic Conditions: A Scoping Review. Nurs Leadersh (Tor Ont). 2019 Sep;32(3):57-76. doi: 10.12927/cjnl.2019.25972. PMID 31714207
- [Background] Gordon K, Dainty KN, Steele Gray C, DeLacy J, Shah A, Seto E. Normalizing Telemonitoring in Nurse-Led Care Models for Complex Chronic Patient Populations: Case Study. JMIR Nurs. 2022 Apr 28;5(1):e36346. doi: 10.2196/36346. PMID 35482375
- [Background] Gordon K, Dainty KN, Steele Gray C, DeLacy J, Shah A, Resnick M, Seto E. Experiences of Complex Patients With Telemonitoring in a Nurse-Led Model of Care: Multimethod Feasibility Study. JMIR Nurs. 2020 Sep 29;3(1):e22118. doi: 10.2196/22118. PMID 34406972
- [Background] Gordon K, Steele Gray C, Dainty KN, DeLacy J, Ware P, Seto E. Exploring an Innovative Care Model and Telemonitoring for the Management of Patients With Complex Chronic Needs: Qualitative Description Study. JMIR Nurs. 2020 Mar 6;3(1):e15691. doi: 10.2196/15691. eCollection 2020 Jan-Dec. PMID 34345777
- [Background] Ware P, Shah A, Ross HJ, Logan AG, Segal P, Cafazzo JA, Szacun-Shimizu K, Resnick M, Vattaparambil T, Seto E. Challenges of Telemonitoring Programs for Complex Chronic Conditions: Randomized Controlled Trial With an Embedded Qualitative Study. J Med Internet Res. 2022 Jan 26;24(1):e31754. doi: 10.2196/31754. PMID 35080502
- [Background] Seto E, Leonard KJ, Cafazzo JA, Barnsley J, Masino C, Ross HJ. Mobile phone-based telemonitoring for heart failure management: a randomized controlled trial. J Med Internet Res. 2012 Feb 16;14(1):e31. doi: 10.2196/jmir.1909. PMID 22356799